CLINICAL TRIAL: NCT02171481
Title: Bioequivalence of Two Different Polymorphs of 150 mg Dabigatran Etexilate Following Oral Administration in Healthy Male and Female Volunteers (Double-blind, Randomised, Single Dose, Replicate Design in a Two Treatments, Four Periods Crossover Phase I Study)
Brief Title: Bioequivalence of Two Different Polymorphs of Dabigatran Etexilate in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1160.66
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

ARMS (2):
- Dabigatran etexilate polymorph II (Experimental)
  Interventions: Drug: Dabigatran etexilate polymorph II
- Dabigatran etexilate polymorph I (Active Comparator)
  Interventions: Drug: Dabigatran etexilate polymorph I

INTERVENTIONS:
Drug: Dabigatran etexilate polymorph II
  Arms: Dabigatran etexilate polymorph II
Drug: Dabigatran etexilate polymorph I
  Arms: Dabigatran etexilate polymorph I

SUMMARY:
To establish the bioequivalence of two polymorphs of dabigatran etexilate, polymorph I and polymorph II

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females according to the following criteria:

   Based upon a complete medical history, including the physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
2. Age ≥60 and ≤85 years
3. BMI ≥18.5 and BMI ≤32.0 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

1. Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Clinically relevant surgery of gastrointestinal tract
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. Any relevant bleeding history
5. History of relevant orthostatic hypotension, fainting spells or blackouts
6. Chronic or relevant acute infections
7. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
8. Intake of drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
10. Participation in another trial with an investigational drug within four weeks prior to administration or during the trial
11. Alcohol abuse (more than 60 g/day for men and more than 40 g/day for women)
12. Drug abuse
13. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
14. Excessive physical activities (within one week prior to administration or during the trial)
15. Any laboratory value outside the reference range that is of clinical relevance
16. Inability to comply with dietary regimen of study centre
17. Planned surgeries within four weeks following the end-of study examination
18. Intake of medication, which influences the blood clotting, i.e., acetylsalicylic acid, coumarin etc. within 10 days prior to administration
19. Male subjects who do not agree to minimise the risk of female partners becoming pregnant from the first dosing day until the completion of the post study medical examination. Acceptable methods of contraception comprises barrier contraception and a medically accepted contraceptive method for the female partner (intra-uterine device with spermicide, hormonal contraceptive since at least two month)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of total BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 72 hours after drug administration
Maximum measured concentration of total BIBR 953 ZW in plasma (Cmax) | Up to 72 hours after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of free BIBR 953 ZW in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 72 hours after drug administration
Maximum measured concentration of free BIBR 953 ZW in plasma (Cmax) | Up to 72 hours after drug administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | Up to 72 hours after drug administration
Area under the concentration time curve of the analyte in plasma over the time interval t1 to t2 with t1 = 0 and t2 = 24, 48, 72 hours (AUCt1-t2) | 24, 48 and 72 hours after drug administration
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | Up to 72 hours after drug administration
Terminal rate constant in plasma (λz) | Up to 72 hours after drug administration
Terminal half-life of the analyte in plasma (t1/2) | Up to 72 hours after drug administration
Mean residence time of the analyte in the body after oral administration (MRTpo) | Up to 72 hours after drug administration
Apparent clearance of the analyte in the plasma after extravascular administration (CL/F) | Up to 72 hours after drug administration
Apparent volume of distribution during the terminal phase λz following an extravascular dose (Vz/F ) | Up to 72 hours after drug administration
Change from baseline in physical examination | Baseline, day 68
Change from baseline in vital signs (blood pressure, pulse rate) | Baseline, day 68
Change from baseline in 12-lead electrocardiogram | Baseline, day 68
Change from baseline in clinical laboratory tests | Baseline, day 68
Number of Participants with Serious and Non-Serious Adverse Events | up to day 68
Assessment of tolerability by investigator on a four point scale (good, satisfactory, not satisfactory, bad) | Day 68